CLINICAL TRIAL: NCT07286617
Title: The Role of Novel STAR Score in Prediction of Intra-Abdominal Injury in Adult Blunt Abdominal Trauma Patients
Brief Title: The Role of Novel STAR Score in Intra-Abdominal Injury in Adult Blunt Abdominal Trauma Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya Mohamed Osman Ali, Resident Physician, Faculty of Medicine - Assiut University, Assiut University
Other Study IDs: STAR-TRAUMA-2025-01
Record Dates: First submitted 2025-09-30; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Novel STAR Score in Prediction of Intra-Abdominal Injury in Adult Blunt Abdominal Trauma Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: STAR Score — The STAR (Screening Tool for Abdominal Injury Risk) score will be applied to adult patients with blunt abdominal trauma to predict intra-abdominal injuries. The score will be calculated based on clinical and laboratory parameters collected at presentation

SUMMARY:
This study aim To develop and assess the diagnostic accuracy of the novel STAR score, combining point-of-care abdominal ultrasound and laboratory parameters, for early prediction of intra-abdominal injuries in adult blunt abdominal trauma patients, and to compare its performance with current standard clinical assessment methods

DETAILED DESCRIPTION:
Blunt abdominal Injury(BAI) can cause damage to Internal organs and internal bleeding. The liver, spleen, and Intestine are the most common organs affected by this type of Injury, and due to the Indirect nature of this injury, diagnosis Is difficult and often time-consuming. Although the outcome of patients with blunt abdominal injury has improved in the last two decades, in patients with multiple organ injuries, the In-hospital mortality rate was reported as 3-10% Early recognition of abdominal trauma is critical, as missed or delayed diagnoses are associated with increased mortality. Clinical assessment, including history, inspection, palpation, percussion, and auscultation, forms the cornerstone of evaluation, but may be limited in accuracy, especially in unconscious or intoxicated patients The development of point-of-care imaging techniques, particularly Focused Assessment with Sonography for Trauma (FAST), has greatly enhanced rapid detection of free intraperitoneal fluid in unstable patients. As a non-invasive, bedside procedure Laboratory investigations play an important adjunctive role in the assessment of abdominal trauma

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 60 years with a documented history of blunt abdominal trauma. Presentation within 6 hours of sustaining the injury.

Hemodynamically stable or unstable patients at the time of presentation:

Stable: Normal blood pressure and heart rate, warm extremities, and capillary refill ≤2 seconds Unstable: Systolic blood pressure <90/60 mmHg or a decrease of >30% from baseline systolic pressure, heart rate >100 beats per minute, cold, clammy skin, and capillary refill time >2 seconds..

Glasgow Coma Scale (GCS) score of 15/15 on initial assessment.

Exclusion Criteria:

* Patients with penetrating abdominal trauma.History of pre-existing abdominal pathology that may interfere with clinical or sonographic assessment (e.g., ascites, prior major abdominal surgery, known masses).

Pregnant patients. Presence of pre-existing infection or hematuria that may alter laboratory parameters.

Patients undergoing cardiopulmonary resuscitation upon arrival. Mechanically ventilated patients at the time of initial assessment.

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Adult patients aged 18-60 years presenting to the Emergency Department with blunt abdominal trauma within 6 hours of injury. Eligible patients include both hemodynamically stable and unstable individuals, provided they have a Glasgow Coma Scale (GCS) of 15/15 at presentation. Patients with penetrating trauma, prior abdominal pathology, pregnancy, infection, hematuria, those requiring cardiopulmonary resuscitation, or on mechanical ventilation at initial assessment will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 129 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2027-11-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Development and validation of a novel ultrasound-laboratory-based scoring system capable of accurately predicting the presence of clinically significant intra-abdominal injury in adult patients with blunt abdominal trauma. | 7 days of admission